CLINICAL TRIAL: NCT05494073
Title: Anterior Cruciate Ligament Reconstruction Hybrid Remnant Repair Randomized Control Trial
Brief Title: Anterior Cruciate Ligament Reconstruction Hybrid Remnant Repair
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Vasilios Moutzouros, Dr. Vasilios Moutzouros M.D. Principle Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14969-01
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Anterior Cruciate Ligament Tear
Keywords: ACL; hybrid remnant repair; Anterior Cruciate Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Remnant Repair (Experimental): Patients in this arm will have an ACL reconstruction with preservation and incorporation of the the ACL remnant.
  Interventions: Procedure: ACL Reconstruction with Hybrid Remnant Repair
- Control (Active Comparator): Patients in this arm will have a ACL reconstruction where the ACL remnant is not incorporated into the graft.
  Interventions: Procedure: ACL Reconstruction without Hybrid Remnant Repair

INTERVENTIONS:
Procedure: ACL Reconstruction with Hybrid Remnant Repair — The intervention includes the incorporation of the host ACL remnant into the graft. The intervention hopefully
  Arms: Hybrid Remnant Repair
Procedure: ACL Reconstruction without Hybrid Remnant Repair — ACL reconstruction without preservation or incorporation of host ACL remnant
  Arms: Control

SUMMARY:
Patients between 14-60 years of age who will undergo an anterior cruciate ligament (ACL) reconstruction between Nov 1, 2021- Dec 31, 2023, will have their charts reviewed be approached in clinic when the surgery is scheduled regarding their participation in this study. At the time of consent, patients will be randomized to a group via a computerized randomization process, either the experimental hybrid remnant repair (HRR) or traditional ACL reconstruction with ACL stump debridement. Routine postoperative data will be collected at regularly scheduled post-operative and physical therapy appointments including range of motion, pain, patient-reported outcomes, return-to-sport tests, and proprioceptive data. Additionally, patients will be asked to undergo a post-operative MRI between 9 and 15 months following the date of their surgery. Radiologists reading the MRIs will be blinded to which group the patient is in. The primary outcome measure is graft incorporation between the two groups.

DETAILED DESCRIPTION:
The purpose of this study is to examine the efficacy of a hybrid remnant repair (HRR) anterior cruciate ligament reconstruction (ACLR) with a traditional ACLR. Orthopedic surgeons are consistently looking for ways to improve outcomes following ACLR. Previous research has focused on different graft harvesting techniques and selection as well as biological augmentation of the graft. Recently, as reconstruction techniques have improved the anatomic accuracy of the reconstruction, there has been a renewed interest in remnant-preserving techniques. Surgeons in the sports medicine department are trained and have been performing HRR for several months at this point. The investigators are interested in comparing the results of patients who underwent HRR ACLR compared to a traditional ACLR.

The specific aim of this investigation is to determine the efficacy of ACL reconstruction with HRR to the standard ACL reconstruction with stump debridement. This study will specifically focus on whether patients who underwent HRR ACLR achieve superior incorporation of the graft, proprioceptive abilities, and improved patient-reported outcomes compared to traditional ACLR. If this procedure provides superior outcomes, it will benefit patients who have an ACL tear with a vascularized remnant stump remaining. The investigators will access information in the Henry Ford electronic medical records and review patient charts to consent patients undergoing ACL reconstruction between June 1, 2021- Dec 31, 2023. The investigators will record intraoperative data including date of surgery, type of graft used, whether or not there was a prior surgery; post-operative data including strength, range of motion, and patient-reported outcomes; all of which are routinely collected or documented. Additionally, between 6 and 15 months postoperatively, patients will undergo postoperative magnetic resonance imaging (MRI) to determine the incorporation of the graft and ACL remnant.

The investigators hypothesize patients undergoing HRR ACLR will have better incorporation with improved vascularity compared to patients undergoing a traditional ACLR. The investigators hypothesize that this will lead to improved proprioceptive abilities and improved patient-reported outcomes, which may reduce the time required to be cleared to return to sport and resume usual activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 14-65 will undergo an anterior cruciate ligament (ACL) reconstruction from June 1,2021-Dec 31,2023 will be chart reviewed and asked about participating in the study in Dr. Moutzouros's clinic at a routine pre-operative clinic appointment .

There will be 100 subjects who are consented, 50 in each group (Arm A- HRR ACLR; Arm B- traditional ACLR with stump debridement).

Exclusion Criteria:

* Patients will be excluded if they suffered concomitant medial collateral ligament (MCL), lateral collateral ligament (LCL), or posterior cruciate ligament (PCL) injury as well as patients who did not undergo HRR ACLR. Additional exclusion criteria includes poor follow-up to post-operative clinic appointments.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Post-operative imaging (MRI) graft incorporation | 1 year post ACLR
  We hypothesize patients undergoing HRR ACLR will have better incorporation with improved vascularity compared to patients undergoing a traditional ACLR. We hypothesize that this will lead to improved proprioceptive abilities and improved patient reported outcomes, which may reduce the time required to be cleared to return-to-sport and resume usual activities of daily living.

SECONDARY OUTCOMES:
Subject proprioceptive ability | Collected at intervals during post-operative period once cleared by physician and physical therapy. 6 weeks, 3 months, 6 months, 12 months since post operative date.
  Patients will be put through a series of tests in line with their clinic visits to objectively test for proprioception. Data will be analyzed and compared between hybrid remnant repair ALCR and traditional ACLR. Tests consist of single leg triple hop for distance and single leg 6 meter hop for time.
Subject quadriceps strength | Collected pre-operatively and at intervals during post-operative period once cleared by physician and physical therapy.6 weeks, 3 months, 6 months, 12 months since post operative date.
  Patients will be subjected to knee extension testing utilizing a dynamometer.
Patient-reported outcomes (PROMIS forms) | Collected pre-operatively and at intervals during post-operative clinic visits. 6 weeks, 3 months, 6 months, 12 months since post operative date.
  Patients will fill out PROM questionnaires in alignment with their clinical visits.
Subject range-of-motion | Collected pre-operatively and at intervals during post-operative clinic visits. 6 weeks, 3 months, 6 months, 12 months since post operative date.
  Range of motion will be assessed with a goniometer.
Return-to-sport (time from surgery) | Variable depending on patients individual recovery. 6 weeks, 3 months, 6 months, 12 months since post operative date.
  Time it takes for patient to return to sport or physical activity formerly participating in prior to ACLR

CONTACTS AND LOCATIONS:
Overall Officials: Vasilios Moutzouros, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
We do not foresee the need to share any individual participant data (IPD) at this time.

REFERENCES:
- [Background] Samuelsen BT, Webster KE, Johnson NR, Hewett TE, Krych AJ. Hamstring Autograft versus Patellar Tendon Autograft for ACL Reconstruction: Is There a Difference in Graft Failure Rate? A Meta-analysis of 47,613 Patients. Clin Orthop Relat Res. 2017 Oct;475(10):2459-2468. doi: 10.1007/s11999-017-5278-9. PMID 28205075
- [Background] Hexter AT, Thangarajah T, Blunn G, Haddad FS. Biological augmentation of graft healing in anterior cruciate ligament reconstruction: a systematic review. Bone Joint J. 2018 Mar 1;100-B(3):271-284. doi: 10.1302/0301-620X.100B3.BJJ-2017-0733.R2. PMID 29589505
- [Background] Tensho K, Iwaasa T, Shimodaira H, Koyama S, Horiuchi H, Takahashi J, Saito N. Anatomical Remnant-Preserving Double-Bundle ACL Reconstruction With a New Remnant Augmentation Technique. Arthrosc Tech. 2020 Jan 24;9(2):e283-e290. doi: 10.1016/j.eats.2019.10.009. eCollection 2020 Feb. PMID 32099783
- [Background] Diaz RMM, Rezende FC, Moscon AC, Franciozi CEDS, Martimbianco ALC, Duarte A. Return to Sports after ACL Reconstruction with Resection or Remnant-Preserving Technique. Rev Bras Ortop (Sao Paulo). 2020 Aug;55(4):432-437. doi: 10.1055/s-0039-3402461. Epub 2020 Feb 7. PMID 32904857